CLINICAL TRIAL: NCT00988234
Title: Comparison of Lateral Decubitus Position Versus Prone Position for Ultrasound Guided Posterior Lumbar Plexus Block and Sciatic Nerve Block
Brief Title: Comparison of Two Position for Ultrasound Guided Lumbar Plexus and Sciatic Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Yuke Tian/ Professor, Department of Anesthesiology, Tongji Hospital, Tongji medical college, Huazhong University of science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJHMZK01001
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Lower Limb Surgery
Keywords: Lumbar plexus block; sciatic nerve block; position; ultrasound guidance; elective lower limb surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SGPP (Experimental): ultrasound guided posterior lumbar plexus block and subgluteal sciatic nerve block under prone position
  Interventions: Procedure: SGPP
- SGTPP (Experimental): ultrasound guided posterior lumbar plexus block and sub-greater trochanter approach under prone position
  Interventions: Procedure: SGTPP
- SGLP (Experimental): ultrasound guided posterior lumbar plexus block and subgluteal sciatic nerve block under lateral decubitus position
  Interventions: Procedure: SGLP
- SGTLP (Experimental): ultrasound guided posterior lumbar plexus block and sub-greater trochanter approach under lateral decubitus position
  Interventions: Procedure: SGTLP

INTERVENTIONS:
Procedure: SGPP — ultrasound guided posterior lumbar plexus block and subgluteal sciatic nerve block under prone position
  Arms: SGPP
Procedure: SGTPP — ultrasound guided posterior lumbar plexus block and sub-greater trochanter approach under prone position
  Arms: SGTPP
Procedure: SGLP — ultrasound guided posterior lumbar plexus block and subgluteal sciatic nerve block under lateral decubitus position
  Arms: SGLP
Procedure: SGTLP — ultrasound guided posterior lumbar plexus block and sub-greater trochanter approach under lateral decubitus position
  Arms: SGTLP

SUMMARY:
In the present study, the investigators will test the effect of two position on posterior lumbar plexus and subgluteal or sub-greater trochanter sciatic nerve block.

DETAILED DESCRIPTION:
The posterior lumbar plexus block approach was described approximately 30 years ago, using surface anatomical landmarks and a loss-of-resistance technique, but over the years it was almost abandoned for its low successful rate, the huge numbers of adverse effects and its difficulties to be performed. The introduction of the nerve stimulator and ultrasound guided technique in recent years increased the success rate in various peripheral nerve blocks and decreased adverse effects. Ultrasound guided LPB as well as sciatic nerve block technique in a small patient population resulting in a encouraging result, but published clinical data on optimal patient position for ultrasound-guided LPB are limited. We designed this prospective randomized study to compare the success rate, time of performance and complications of ultrasound guided posterior lumbar plexus block as well as subgluteal or sub-greater trochanter sciatic nerve block under lateral decubitus position v.s. prone position.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* elective unilateral lower limb surgery
* ASA Physical Status ASA I-III

Exclusion Criteria:

* age <18 or >75 year old
* ASA Physical Status >ASA III
* abnormal blood coagulation
* infection near puncture place
* nerve injury
* bilateral lower limb surgery
* patients with lumbar vertebral trauma
* inability to be properly positioned
* chronic narcotic therapy or illicit drug use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Block success defined as loss of sensation to pinprick in each of the lumbar plexus and sciatic nerve distributions when measured 30 min after block performance. | 30min
Motor blockade was evaluated by assessing the strength of knee extension (femoral nerve), thigh adduction (obturator nerve), and plantar flexion and dorsiflexion of the ankle (sciatic nerve) 30 min after block performance. | 30min

SECONDARY OUTCOMES:
block execution time, depth of the nerve, needle depth, duration of the sensory and motor blockade, complications such as inadvertent needle puncture of epidural space, dural puncture, peritoneal puncture, and kidney or ureter puncture and nerve injury. | within 48h

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, MD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China